CLINICAL TRIAL: NCT02887885
Title: Sustainability of Vaginal Estrogen Therapy in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Medinova AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-00380
Record Dates: First submitted 2016-08-17; First posted 2016-09-02 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Atrophy of Vagina; Postmenopause

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gynoflor — 1 vaginal tablet daily for 12 days, followed by 3 vaginal tablets per week as maintenance therapy (Monday-Wednesday-Friday) for 6 weeks

SUMMARY:
Sustainability of vaginal ultra-low dose estrogen therapy in postmenopausal women

DETAILED DESCRIPTION:
Within this trial 50 postmenopausal women receive a vaginal estrogen therapy as treatment for symptomatic vaginal atrophy. The sustainability of vaginal estrogen therapy after the end of therapy has not yet been investigated.

All participants will be asked to come for the following 7 visits.

* Visit 1: Standard Gynecological examination; Inclusion and exclusion criteria check
* Visit 2: Handing out of Gynoflor (estrogen) for a 6 weeks treatment.
* Visit 3 (Study Start): After using the vaginal estrogen for 6 weeks, a vaginal swap will be done to measure the vaginal maturation index (VMI). The participants will also receive a questionnaire to define some subjective parameters. The parameters measured at visit 1 will count as reference. The estrogen therapy will now be sustained.
* Visit 4-6: Measuring of the VMI and handing out the questionnaires to define subjective parameters.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (last menstrual period more than 12 months ago or having undergone bilateral ovariectomy)
* Age ≥ 18 years
* Diagnosis of moderate to severe vaginal atrophy at screening visit with VMI < 50% and vaginal pH > 4.5
* At least one subjective symptom of vaginal atrophy (dryness, pain/burning sensation, pruritus, discharge, dyspareunia) related to a score of ≥ 65 on the visual analogue scale (VAS)
* Indication for vaginal treatment with Gynoflor® (100 million viable L. acidophilus KS 400 and estriol 30 mcg per application) for 6 weeks because of symptomatic vaginal atrophy after menopause: 1 vaginal tablet daily for 12 days, followed by 3 vaginal tablets per week as maintenance therapy (Monday-Wednesday-Friday).
* Informed consent as documented by signature

Exclusion Criteria:

* Administration of any form of oral/transdermal hormone therapy (HT) or selective estrogen receptor modulators (SERM) or phytoestrogens within 2 months prior to entry into or during the study.
* Any use of over-the-counter vaginal products within 1 week prior to and during entry the study.
* Known hypersensitivity or allergy to the investigational product
* Estrogen dependent malignancy
* Undiagnosed genital bleeding
* Active thromboembolism
* Active vulvovaginal Candidiasis, Trichomonas vaginitis or bacterial vaginitis based on light microscopy of vaginal secretions, vaginal pH, whiff test and KOH preparation
* Active sexually transmitted infections (STI) including herpes simplex viral infection, gonorrhoea and Chlamydia.
* Active urinary tract infection.
* Pessary-users
* Immunocompromised patients including those with human immunodeficiency viral infection, chronic glucocorticoid use or active treatment with immunosuppressive agents
* Severe liver and/or kidney disease
* Diabetes mellitus
* Polyneuropathy
* Skin disease affecting vulva or vagina, e.g. lichen sclerosus
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Mean change in vaginal maturation index (VMI) | 0 weeks, 4 weeks

SECONDARY OUTCOMES:
Mean change in VMI | 0 weeks,1 week, 2 weeks, 6 weeks
Mean change in vaginal pH | 0 weeks,1 week, 2 weeks, 4 weeks, 6 weeks
Number of lactobacilli | 0 weeks,1 week, 2 weeks, 4 weeks, 6 weeks
Lactobacillary grade (LBG), | 0 weeks,1 week, 2 weeks, 4 weeks, 6 weeks
Mean change in the most bothersome moderate and severe symptom of vaginal atrophy (MBS) . The symptoms include dryness, pain/burning sensation, pruritus, discharge, and dyspareunia. | 0 weeks,1 week, 2 weeks, 4 weeks, 6 weeks
Mean change in health-related quality of life (EQ-5D-5L). Mean change in Female Sexual Function Index (FSFI). | 0 weeks,1 week, 2 weeks, 4 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, Prof, Principal Investigator — University Hospital Berne
Locations (1):
- Dep. of Obstetrics and Gynecology, Bern University Hospital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562
- [Background] McEndree B. Clinical application of the vaginal maturation index. Nurse Pract. 1999 Sep;24(9):48, 51-2, 55-6. PMID 10507070